CLINICAL TRIAL: NCT00137332
Title: A Study of the Effects GAP-486 on Ventricular Tachyarrhythmia Induction
Brief Title: Study Evaluating GAP-486 on Heart Rhythm in Patients With Coronary Artery Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3163K1-202
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2007-12-10 (Estimated); Status verified 2007-12

CONDITIONS: Arrhythmia
Keywords: Arrhythmia; antiarrhythmic; programmed electrical stimulation
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — rotigaptide; Sodium Chloride

INTERVENTIONS:
Drug: GAP-486 (ZP-123)
Drug: 0.9% Sodium Chloride, USP

SUMMARY:
The purpose of this study is to learn the effects of a test drug on heart rhythms, which may become life-threatening if left untreated, and to provide data to see if the drug is well tolerated and safe.

ELIGIBILITY:
Inclusion Criteria:

* Patients with or without ICDs (implantable cardioverter defibrillators)
* Patients undergoing an electrophysiology study for evaluation of ventricular rhythm
* Patients with a history of heart disease

Exclusion Criteria:

* Patients with uncontrolled blood pressure
* Patients with certain cardiac risk factors
* Patients with significant kidney or liver problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2005-11; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The measure to determine the effect of the intervention will be whether abnormally fast heart rhythm can be induced after test drug is administered.

SECONDARY OUTCOMES:
This study takes place within 24 hours, and looks at whether the test article makes a difference in inducing the abnormally fast heart rhythm during a 24 hour observational period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (30):
- United States (18):
  - Sacramento, California
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Orlando, Florida
  - Peoria, Illinois
  - Iowa City, Iowa
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Lansing, Michigan
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Newark, New Jersey
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Wynnewood, Pennsylvania
  - Falls Church, Virginia
  - Norfolk, Virginia
- Canada (12):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - St-Johnâ S, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - London, Ontario
  - Newmarket, Ontario
  - Toronto, Ontario
  - Fleurimont, Quebec
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec